CLINICAL TRIAL: NCT01597362
Title: Three Laparoscopic Access Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Cafa Ester Valentina, Principal Investigator, Campus Bio-Medico University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TRC-01
Record Dates: First submitted 2012-05-09; First posted 2012-05-14 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Benign Gynecological Pathology
Keywords: laparoscopy; trocars; veress; open; direct
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Veress needle technique (Other)
  Interventions: Procedure: Laparoscopy
- Direct trocar technique (Other)
  Interventions: Procedure: Laparoscopy
- Open technique (Other)
  Interventions: Procedure: laparoscopy

INTERVENTIONS:
Procedure: laparoscopy — Trocar access in laparoscopy
  Arms: Open technique
Procedure: Laparoscopy — The angle of the Veress needle insertion is 45 for non-obese women. After insertion of the needle, tests to determinate its correct positioning are: the double click test, the aspiration test, the handing drop test, serial intrabdominal gas pressure measurements.
  The volume of CO2 inserted with the Veress needle depends on the intra-abdominal pressure. Adequate pneumoperitoneum should is determined by a pressure of 20 to 30 mm Hg and not by predetermined CO2 volume.
  Arms: Veress needle technique
Procedure: Laparoscopy — Direct insertion of the trocar is performed without prior pneumoperitoneum. Infra-umbilical skin incision is wide enough to accomodate the diameter of a sharp trocar/cannual system. The abdominal wall is elevated by pulling on, by hands, two towel clips placed 3 cm on either side of the umbilicus, and the trocar is inserted at a 90°angle.
  On removal of the sharp trocar, the laparoscope is inserted to confirm the presence of omentum or bowel in the visual field.
  Arms: Direct trocar technique
Procedure: Laparoscopy — A small incision, 1 cm long, is made through the skin of the lower edge of the umbilical fossa. The skin and the subcutaneous adipose tissues are retracted with the Zimmerman dissectors. The anterior rectus fascia is incised with the scalpel. The dissection with the Zimmerman valves allows the exposure of the peritoneum. After the peritoneum is incised, the trocar is inserted under direct vision. The laparoscope is introduced and insufflation is started. At the end of the procedure the fascial defect is closed.
  Arms: Open technique

SUMMARY:
The study compares the Veress needle technique, the Direct trocar insertion and the Open technique with each other, in terms of minor complications, in elective laparoscopic procedures for benign pathologies.

ELIGIBILITY:
Inclusion Criteria:

* not-obese adult patients referred for scheduled laparoscopic and gynecologic procedures,
* benign pathology
* no previous abdominal surgery
* Age range was 18-70 years

Exclusion Criteria:

* obesity, defined as a body mass index (BMI) > 30 kg/m2
* previous abdominal surgery by laparoscopy or laparotomy
* history of PID
* irritable Bowel Syndrome
* suspicion of malignancy or malignancy at the histological examination

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2006-02; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
minor complications | 1 year
  feasibility of the techniques and the incidence of Veress needle, Direct technique insertion and Open technique related minor complications

REFERENCES:
- [Derived] Angioli R, Terranova C, De Cicco Nardone C, Cafa EV, Damiani P, Portuesi R, Muzii L, Plotti F, Zullo MA, Panici PB. A comparison of three different entry techniques in gynecological laparoscopic surgery: a randomized prospective trial. Eur J Obstet Gynecol Reprod Biol. 2013 Dec;171(2):339-42. doi: 10.1016/j.ejogrb.2013.09.012. Epub 2013 Sep 23. PMID 24103531